CLINICAL TRIAL: NCT00355433
Title: Comparison of Urodynamic Volume Measurements Using Room and Body Temperature Saline
Brief Title: Comparison of Body and Room Temperature Saline in Urodynamics
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tripler Army Medical Center (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Diagnostic
Other Study IDs: TAMC 11H06
Record Dates: First submitted 2006-07-20; First posted 2006-07-24 (Estimated); Last update posted 2006-07-24 (Estimated); Status verified 2006-07

CONDITIONS: Urinary Incontinence
Keywords: urinary incontinence; urodynamics; temperature
MeSH Terms: conditions — Urinary Incontinence

INTERVENTIONS:
Procedure: Urodymanics

SUMMARY:
The purpose of this study is to compare first urge, strong urge, and maximum capacity, and perception of discomfort during urodynamic testing between room temperature and body temperate saline. Twenty-four non-pregnant females referred to the urogynecology clinic for bladder testing will be enrolled into the study. Each patient will serve as her own control, undergoing the bladder testing with both room temperature and body temperature saline.

DETAILED DESCRIPTION:
This is a prospective observational study. Patient scheduled to undergo evaluation of urinary incontinence by urodynamics in the gynecology clinic will be asked to participate. Patients will be counseled and consent forms signed. The nurse will open the envelope which randomizes the order of instillation and set up the first fluid. Normal saline in 1000ml bags are used for instillation. The bags being used for body temperature fluid will be heated using an Olympic Warmette to between 98 and 99 degrees as determined by 3M Tempadot Thermometers. Urodynamics will be performed using standard clinic protocol recording first sensation, first urge, and maximum capacity. The patient will ask to comment on the discomfort of the test using a 5 point Lickert scale for both pain and urgency (see attached questions). Patients will be allowed to void. The bladder will be filled again with the second solution with identical questions used to determine first sensation, first urge and maximum capacity. During each filling the patient will be tested for stress incontinence at 200 and 300 mls as per our protocol. Following the instillation of the second solution the patient will again be asked her perception of pain and urgency an identical scale. Maximum bladder capacities from each temperature saline tested will then be compared against maximum bladder capacity as estimated from the patients' bladder diary. The patient will then be managed as is appropriate for her test results.

ELIGIBILITY:
Inclusion Criteria:

* Females referred to gynecology clinic for urodynamics evaluation with an appropriate indication for bladder testing

Exclusion Criteria:

* Male subjects and pregnant females

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24
Dates: Start 2006-07; Study Completion 2006-07

PRIMARY OUTCOMES:
first urge
strong urge
maximum urge

SECONDARY OUTCOMES:
patient comfort (Likert scale)

CONTACTS AND LOCATIONS:
Locations (1):
- Tripler Army Medical Center, TAMC, Hawaii, United States

REFERENCES:
- [Background] 1. Klevmark, B, Volume threshold for micturation: Influence of filing rate on sensory and motor bladder function, Scandanavian Journal of Urology and Nephrology Supplementum 2002; 210:6-10 2. Wyandaele, J, The normal pattern of perception of bladder filling during cystometry studied in 38 young healthy volunteers, Journal of Urology 1998; 160(2):479-81 3. Pauwels, E, DeWatcher, S, Wyndaele, J, Normality of bladder filling studied in symptom-free middle-aged woman, Clinical Urology 2004; 171(4):1567-70 4. Chin-peuckert, L, Komlos, M, Rennick, J, Jednak, R, Capolicchio, J, Salle, J, What is the variability between two concescutive cystometries in the same child?, Clinical Urology 2003; 170(4):1614-7 5. Goodman, T, Kilborn, T, Pearce, R. Warm or cold contrast medium in the micturating cystourethrogram: which is best?, Clinical Radiology 2003; 58(7):551-4